CLINICAL TRIAL: NCT02189577
Title: A Multinational, Multicentre, Randomised, Double Blind, Placebo-Controlled, 2-way Crossover Study to Evaluate the Efficacy and Safety of Glycopyrrolate Bromide Administered Via pMDI (CHF 5259), for the Treatment of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Glycopyrrolate Bromide of COPD Patients
Acronym: Trigon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-05993AA1-09; 2013-005268-25 (EudraCT Number)
Record Dates: First submitted 2014-07-02; First posted 2014-07-14 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 5259 (Experimental): CHF 5259
  Interventions: Drug: CHF 5259
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF 5259 — Comparison of CHF 5259 versus placebo over a treatment period. Allocation of 1 of the 2 possible treatments performed in sequence during a cross over design.
  Other Names: glycopyrrolate bromide
  Arms: CHF 5259
Drug: Placebo — Comparison of CHF 5259 versus placebo over a treatment period. Allocation of 1 of the 2 possible treatments performed in sequence during a cross over design.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CHF 5259 (glycopyrrolate bromide) for the treatment of COPD patients.

DETAILED DESCRIPTION:
A Multinational, Multicentre, Randomised, Double Blind, Placebo-Controlled, 2-way Crossover Study to Evaluate the Efficacy and Safety of Glycopyrrolate Bromide Administered Via pMDI (CHF 5259), for the Treatment of Patients With Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (40 ≤ age ≤ 80 years) with a diagnosis of COPD
* Current smokers or ex-smokers
* A post-bronchodilator FEV1 < 60% of the predicted normal value and a post-bronchodilator FEV1/FVC < 0.7
* Positive response to the reversibility test at screening defined as change in FEV1 ≥ 5%.
* BDI score ≤ 10
* Patients free of exacerbations for at least 1 month

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of asthma
* Patients treated for exacerbations in the 4 weeks prior to screening visit
* Patients treated with long-acting antihistamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study or if taken as PRN
* Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia
* Known respiratory disorders other than COPD
* Patients who have clinically significant cardiovascular condition

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pre-dose morning FEV1 on Day 28 | Day 28

SECONDARY OUTCOMES:
Change from baseline to day 28 in area under the curve for forced expiratory volume in 1 second measured at 11 timepoints between 0 to 12 hours postdose (FEV1 AUC0-12h) | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Michael POLKEY, MD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust; South Kensington Campus, London SW7 2AZ; UK
Locations (29):
- Bulgaria (8):
  - Chiesi Clinical Trial Site 1017, Sevlievo
  - Chiesi Clinical Trial Site 1010, Sofia
  - Chiesi Clinical Trial Site 1011, Sofia
  - Chiesi Clinical Trial Site 1014, Sofia
  - Chiesi Clinical Trial Site 1015, Sofia
  - Chiesi Clinical Trial Site 1016, Sofia
  - Chiesi Clinical Trial Site 1012, Stara Zagora
  - Chiesi Clinical Trial Site 1013, Troyan Municipality
- Germany (8):
  - Chiesi Clinical Trial Site 2024, Berlin
  - Chiesi Clinical Trial Site 2028, Berlin
  - Site 2020 - Pulmonary Research Institute at Hospital Grosshansdorf, Großhansdorf
  - Chiesi Clinical Trial Site 2027, Hamburg
  - Chiesi Clinical Trial Site 2026, Leipzig
  - Chiesi Clinical Trial Site 2023, Magdeburg
  - Chiesi Clinical Trial Site 2021, Radebeul
  - Chiesi Clinical Trial Site 2022, Witten
- Poland (10):
  - Chiesi Clinical Trial Site 3039, Bydgoszcz
  - Chiesi Clinical Trial Site 3032, Katowice
  - Chiesi Clinical Trial Site 3035, Krakow
  - Chiesi Clinical Trial Site 3037, Lubin
  - Chiesi Clinical Trial Site 3031, Ostrowiec Świętokrzyski
  - Chiesi Clinical Trial Site 3033, Oświęcim
  - Chiesi Clinical Trial Site 3038, Rzeszów
  - Chiesi Clinical Trial Site 3034, Tarnów
  - Chiesi Clinical Trial Site 3030, Wroclaw
  - Chiesi Clinical Trial Site 3036, Zgierz
- United Kingdom (3):
  - Site 4040 - Royal Brompton and Harefield NHS Foundation Trust; South Kensington Campus, London
  - Chiesi Clinical Trial Site 4042, London
  - Chiesi Clinical Trial Site 4041, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2013-005268-25
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-05993AA1-09.pdf